CLINICAL TRIAL: NCT03199586
Title: First-in-Human, Dose Finding, Open Label Phase 1A-1B Clinical Trial of Metastasis Inhibitor NP-G2-044 in Patients With Advanced or Metastatic Treatment-Refractory Solid Tumor Malignancies
Brief Title: Clinical Trial of Metastasis Inhibitor NP-G2-044 in Patients With Advanced or Metastatic Treatment-Refractory Solid Tumor Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novita Pharmaceuticals, Inc. (Industry)
Collaborators: Translational Drug Development (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP-G2-044-P1-01
Record Dates: First submitted 2017-06-23; First posted 2017-06-27 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer; Pancreas Cancer; Prostate Cancer; Lung Cancer; Colon Cancer; Esophagus Cancer; Liver Cancer; Ovary Cancer; Advanced or Metastatic Treatment-refractory Solid Tumor Malignancies
Keywords: Advanced or metastatic treatment-refractory solid tumor malignancies
MeSH Terms: conditions — Breast Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms; Lung Neoplasms; Colonic Neoplasms; Esophageal Neoplasms; Liver Neoplasms; Ovarian Neoplasms | interventions — NP-G2-044

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NP-G2-044 (Experimental): capsule
  Interventions: Drug: NP-G2-044

INTERVENTIONS:
Drug: NP-G2-044 — capsule

SUMMARY:
Phase 1 A: First-in-human phase 1 study to determine safety of NP-G2-044 when given orally on a daily X 28 days followed by a 14 day rest period.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent and mental capability to understand the informed consent
2. Male or female patients > 18 years of age
3. Histologically or cytologically documented locally advanced or metastatic solid tumor malignancies either treatment-refractory or otherwise ineligible for treatment with standard-of-care agents/regimens
4. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1
5. Evaluable or measurable disease per RECIST v1.1
6. Life expectancy > 3 months
7. ECG without evidence of clinically meaningful conduction abnormalities or active ischemia as determined by the Investigator
8. Acceptable organ and marrow function as defined below:

   * Absolute neutrophil count > 1,500 cells/μL
   * Hemoglobin ≥ 9.0 g/dL
   * Platelets > 100,000 cells/μL
   * Total bilirubin ≤ 1.5 mg/dL
   * Albumin ≥ 3 g/dL
   * Aspartate aminotransferase (AST)/alanine transaminase (ALT)/alkaline phosphatase (ALP)/Gamm-glutamyl transferase (GGT) ≤ 2.5 times ULN. For Phase 1A only, if liver metastases are present, AST/ALT/ALP < 5 times ULN
   * Serum creatinine < 1.5 mg./dL and a measured creatinine clearance ≥ 60 mL/min
   * Prothrombin time (PT)/partial thromboplastin time (PTT) ≤ 1.5 times ULN
9. Women of child-bearing potential (defined as a female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or is not postmenopausal (defined as amenorrhea for at least 12 consecutive months with an appropriate clinical profile at the appropriate age, e.g., greater than 45 years) must have a negative serum pregnancy test prior to first dose of study drug.
10. Male and female patients with reproductive potential must agree to use adequate contraceptive precautions throughout the study.

Exclusion Criteria:

1. Chemotherapy, radiotherapy or other anti-cancer treatment within 4 weeks or 5 half-lives (whichever is shorter) (6 weeks for nitrosoureas or mitomycin C) of the first dose of study drug or patients who in opinion of Investigator have not recovered from AEs due to agents administered greater than 4 weeks earlier (prior immunotherapy is allowed)
2. Participation in any other clinical investigation using an experimental drug within 4 weeks of first dose of study drug
3. Failure to recover to ≤ grade 1 toxicity (except grade 1-2 alopecia or neuropathy) associated with previous chemotherapy, radiotherapy, biologic, hormone or prior investigational therapy
4. Known untreated brain metastases or treated brain metastases that have not been radiographically and clinically stable (i.e. not requiring steroids) ≥ 4 weeks prior to study enrollment
5. Baseline prolongation of QT/QTc interval (QTc interval > 470 msec in women and >450 msec in men)
6. Uncontrolled intercurrent illness (including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations) that in opinion of Investigator would limit compliance with study requirements
7. Women who are pregnant or breastfeeding
8. Prior allogenic hematopoietic stem cell transplant or allogenic bone marrow transplant or prior solid organ transplant or current use of immuno suppression drugs or anti-transplant rejection drugs
9. Prior history of clinically significant gastrointestinal bleeding, intestinal obstruction or gastrointestinal perforation within 6 months of study enrollment
10. Sponsor reserves right to exclude any patient from the study on basis of pre-study medical histories, physical examination findings, clinical laboratory results, prior medications, or other entrance criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2020-05-07 (Actual)

PRIMARY OUTCOMES:
Establish the safe recommended phase 2 dose | 24 months
  Treatment related adverse events assessed by CTCAE V4.03

SECONDARY OUTCOMES:
Identify and characterize preliminary anti tumor activity | 24 months
  Anti tumor activity assessed using RECIST 1.1
Characterize the pharmacokinetics of NP-G2-044 | 24 months
  Drug exposure assessed by area under the curve (AUC)
Tmax | 24 months
  Time to peak plasma concentration
Cmax | 24 months
  Peak plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Jillian Zhang, Ph.D., Study Director — Novita Pharmaceuticals
Locations (3):
- United States (3):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - City of Hope National Medical Center, Duarte, California
  - Memorial Sloan Kettering Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sever S. Role of actin cytoskeleton in podocytes. Pediatr Nephrol. 2021 Sep;36(9):2607-2614. doi: 10.1007/s00467-020-04812-z. Epub 2020 Nov 13. PMID 33188449